CLINICAL TRIAL: NCT01151969
Title: Effectiveness of the "7H" Intervention to Reduce Frequent Attendance in Primary Care: Cluster Randomised Controlled Trial. The "7H" Study
Brief Title: Effectiveness of the "7H" Intervention to Reduce Frequent Attendance in Primary Care
Acronym: "7H"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mediterranean Institute for the Advance of Biotechnology and Health Research (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Juan Ángel Bellón Saameño, PhD Medicine, The Mediterranean Institute for the Advance of Biotechnology and Health Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PI-0505
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Frequent Attenders
Keywords: Health Service Misuse; Overutilization of Health Services; Primary Health Care; Cost Effectiveness; Quality of life; Randomised Controlled Trial; Multilevel analysis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New multicomponent intervention (Experimental)
  Interventions: Behavioral: New multicomponent "7H" intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: New multicomponent "7H" intervention — The GPs in the intervention group will undertake an interactive workshop training session (15 hours) on the '7 hypotheses' (7H) intervention. In short, this intervention encourages GPs to select from a list of seven possible hypotheses for why the patient is a frequent attender: biological, psychological, social, family, cultural, administrative-organisational, or related to the doctor-patient relationship.
  Arms: New multicomponent intervention

SUMMARY:
The main objective is to measure the effectiveness of a new intervention to decrease use of services of primary care frequent attenders (FA).Among the secondary objectives are to evaluate the cost-effectiveness and cost utility of the new intervention compared with usual care.

METHODS: There will be a randomized controlled trial with cluster assignment. It will take place in the field of primary care in the city of Malaga.It will be evaluated a new multicomponent intervention called "7H" (7 Hypothesis). This intervention will be applied on the FA by their family doctors in the intervention group. In the control group will be developed usual cares.

The main outcome is the total of visits of FA at 12 months of the follow-up. The secondary outcomes include changes happened in biopsychosocial health, satisfaction, and quality of life measurements. The investigators will assess the dependent and independents (from FA, general practitioner [GP] and health centres) variables at baseline, and 12 months. At baseline it will be include a random sample of 450 FA (225 for each arm), belonging to 30 family doctors of 10 health centres. It will be performed linear regression multilevel models with 4 levels (time, patient, doctor and health centre) to evaluate the effectiveness of the intervention. . Moreover will be undertaken multivariate gamma and quantile regressions to assess the cost-effectiveness and cost-utility respectively of the new intervention versus usual cares, estimating their standard errors by bootstrap calculations.

DETAILED DESCRIPTION:
The "7H" intervention

1. Hypothesis generation: analysis of available informationGPs analyze all the available information about possible reasons for frequent attendance from clinical charts using a standardized questionnaire designed to facilitate analysis of this information. This questionnaire prompts analysis of the following: (1) category of visits and their frequencies; (2) type of frequent attender according to the first point; (3) family and personal history, and biopsychosocial problem list that needed follow-up; (4) searching for common factors for frequent attendance from the previous points; (5) feelings and thoughts questionnaires, 'In most interviews with this patient I think ...' (11 items), 'I feel ...' (13 items); (6) rethinking issues of GP capacity (and processes) to resolve the frequent attendance in this patient; and (7) analyzing the different professionals who intervened in patient care and their contribution to resolving or continuing frequent attendance.Finally, GPs indicate the type of hypothesis from a list of seven that they believe made the patient a frequent attender: biological, psychological, social, family, cultural, administrative-organizational, or related to the doctor-patient relationship.
2. Hypothesis confirmation: the decision to accept or refute each hypothesis is based on the GP's interpretation of the data (cognitive component) and the self-perception about feeling sure (emotional component). When necessary, the GPs can try out the hypothesis with one or more of the following strategies: another interview with the patient,biological and psychosocial tests, and/or asking for the opinion of other professionals.
3. Planning: the GP makes plans for each frequent attender based on the confirmed hypothesis and available resources. There are many possible plans, examples of which include: making longer intervals between medical revisits for stable chronic patients, and asking for collaboration with nurses; looking for possible causes of the unstable physical chronic illness and intervening accordingly; scheduling an interview to search for a psychological, family or/and, social diagnosis; suppressing unnecessary face-to-face medical revisits for repeat prescriptions in stable chronic patients, and asking the health centre administrative staff for collaboration; asking the social worker at the health centre for help; referring to community resources if necessary; and being more realistic about the type of doctor-patient relationship expected. These plans are then commented on at the group meeting, after which the GP negotiates the plan with the frequent attender. The GP should never suggest to the patient: 'You have to attend less frequently'. This would be too aggressive and the patient might react with anger or guilt. It is better to offer a search for solutions to the patient's health problem from both points of view.

ELIGIBILITY:
Inclusion Criteria:

* Frequent Attenders: 90th percentile of number of visits of the previous year, stratified by age and sex.

Exclusion Criteria:

* < 14 years.
* Unable to understand or speak Spanish.
* Cognitive impairment.
* Terminal illness.
* Planning to be outside of the the city 3 or more months during the next 12 months.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the intervention "7H" | 12 months

SECONDARY OUTCOMES:
Cost-effectiveness and cost-utility | 12 months
  To evaluate the cost-effectiveness and cost-utility of the intervention "7H" versus usual care.

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio Andaluz de Salud. Distrito Sanitario Málaga, Málaga, Málaga, Spain